CLINICAL TRIAL: NCT00006262
Title: A Phase 2 Study of BMY-27557-14 (a Rebeccamycin Analog) in Patients With Ovarian Cancer
Brief Title: Rebeccamycin Analogue in Treating Patients With Refractory Stage III or Stage IV Ovarian Epithelial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to accrue patients to the study.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NCI 00G1; NU-NCI-00G1; NCI-1132
Record Dates: First submitted 2000-09-11; First posted 2004-03-25 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Ovarian Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — becatecarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: becatecarin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of rebeccamycin analogue in treating patients who have refractory stage III or stage IV ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate to rebeccamycin analogue in patients with refractory stage III or IV ovarian epithelial cancer who have failed platinum in combination with paclitaxel chemotherapy. II. Determine the toxicities of this treatment regimen in these patients.

OUTLINE: Patients receive rebeccamycin analogue IV over 60 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients with complete response after receiving 3 courses receive 3-6 additional courses. Patients with partial response or stable disease after receiving 3 courses receive 3-12 additional courses. Patients with complete response are followed every 2 months for 2 years, and then every 3 months thereafter. All other patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 18-39 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed stage III or IV ovarian epithelial cancer Platinum resistant disease as defined by disease progression during or within 6 months of receiving prior paclitaxel combined with cisplatin or carboplatin No elevated CA-125 as only evidence of disease recurrence Measurable disease At least 20 mm in diameter by conventional techniques OR At least 10 mm in diameter by spiral CT scan No known brain metastases

PATIENT CHARACTERISTICS: Age: 21 and over Performance status: ECOG 0-2 Life expectancy: Greater than 3 months Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal AST and ALT no greater than 2.5 times upper limit of normal Renal: Creatinine normal OR Creatinine clearance greater than 60 mL/min Other: No history of allergic reactions to compounds of similar chemical or biologic composition to rebeccamycin analogue No other prior cancer within the past 5 years except nonmelanomatous skin cancer No other medical problems that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: No other concurrent therapeutic agents for cancer

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-07; Primary Completion 2001-09 (Actual); Study Completion 2001-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Fishman, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States